CLINICAL TRIAL: NCT03915002
Title: Integrated Approaches for Identifying Molecular Targets in Liver Disease
Acronym: InLi
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Gavin Arteel, Professor, University of Pittsburgh
Other Study IDs: STUDY19120198
Record Dates: First submitted 2019-04-05; First posted 2019-04-16 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Alcoholic Liver Disease; Non-Alcoholic Fatty Liver Disease; Steatohepatitis, Nonalcoholic; Steatohepatitis
MeSH Terms: conditions — Liver Diseases, Alcoholic; Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — -Serum, plasma, whole blood, urine, stool, liver tissue, visceral fat and saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients: Steatohepatitis:
  1. Alcoholic Steatohepatitis and Alcoholic liver disease
  2. Nonalcoholic fatty liver disease (NAFLD) and Nonalcoholic Steatohepatitis (NASH)
- Disease control: Patients 18 years or older with a diagnosis of cholestatic liver diseases (primary biliary cholangitis or primary sclerosing cholangitis) or hepatotropic virus (hepatitis C or B virus), according to the current international guidelines.
- Control subjects: Patients over 18 years old without a diagnosis of liver disease that for any other reason (i.e candidate to liver donor, patients with liver metastasis that require surgery, patients with any type of benign liver tumor or HCC in a healthy liver).
  Patient over 18 years old with a documented alcoholic used disorder in their clinical records and without any evidence of liver disease.

SUMMARY:
To provide a framework for successful clinical trials testing novel targets for therapy in liver disease.

To identify molecular and cellular drivers of liver disease to provide a molecular classification and study the determinants or key drivers of disease progression.

Consecutive patients admitted with steatohepatitis (alcoholic or non-alcoholic) will be enrolled in this study where liver tissue, blood and stool will be collected to discover and validate factors associated with diagnosis, severity, histological characteristics, development of decompensations, progression of disease and survival.

DETAILED DESCRIPTION:
In 2015, chronic liver diseases were responsible for approximately 2% of worldwide mortality and in 2016 cirrhosis and chronic liver diseases accounted for 531.1 age- standardized, Disability Adjusted Life Years (DALY's) /100,000 habitants.(1, 2) Cirrhosis is a leading cause of death worldwide within adults between 50 and 70 years old. In the past few decades vast improvements have been made, death rates have decreased for almost all diseases. However, in the USA, the occurrence of alcoholic cirrhosis and HCV cirrhosis has increased, 79 and 75% respectively, from 1990 to 2016 in regards of total number of deaths (3). This trend can also be observed in other countries such as UK where standardized mortality rates have increased 400% in the last 44 years. This has a big impact in the working-age population (18-65 years old)(4). The main causes of liver cirrhosis are hepatitis B virus (HBV) and C (HCV) as well as alcoholic and non-alcoholic fatty liver disease (ALD and NAFLD, respectively).

Most chronic liver diseases have a silent course until the development of complications. For patients with compensated disease, the presence of significant liver fibrosis predicts decompensated disease and early mortality.(5-8) Therefore, diagnosis at early stages is mandatory to prevent liver-related morbidity and mortality.

The aim of this project is to provide a framework for successful clinical trials testing novel targets for therapy in liver disease. The "Integrated Approaches for Identifying Molecular Targets in Liver Disease" (InLi) group is aimed to fill this gap. The group InLi will be composed of a multidisciplinary group including hepatologists, physician-scientists, basic scientists and bioinformatics experts. The main goal of InLi is to provide a framework for successful clinical trials testing novel targets for therapy in alcoholic hepatitis. The Human Biorepository Core will include a variety of biological samples from patients with a wide arrange of liver diseases as well as healthy controls from UPMC liver center as well as a comprehensive database that includes epidemiological, dietary, anthropometrical, analytical, histological, and clinical data.

A common protocol for tissue processing, shipping and storage will be used to ensure sample integrity and quality. Storage of data generated from patients and biospecimens will be facilitated through, Research Electronic Data Capture (REDCap) system, and will follow strict security measures including encryption, coding and limited access to the database.

The development of new-targeted therapies for most liver diseases, but especially, steatohepatitis, one of the more urgent needs in clinical hepatology. To reach this goal, a large multidisciplinary network is required. InLI coordinates a multidisciplinary group composed of clinicians, physician-scientists, basic scientists and bioinformatics experts. The overarching hypothesis of InLi is that the most rational way to provide a useful framework for future clinical trials in liver disease consists of the (i) determination of key drivers of the disease process, (ii) classification of molecular profiles and subtypes of specific liver diseases within each and every pathology, and (iii)identification of "druggable" targets based on both key drivers and molecular classification.

The Human Biorepository Core will generate a large collection of samples from patients with different Liver diseases (e.g. viral, steatohepatitis and cholestasis liver disease). For each disease, we will consider a range of phenotypes focusing in early, intermediate and late disease stages and for each etiology. Moreover, we will also include samples from control patients. We will also build a comprehensive database that will serve as a basis for the proposed translational studies and be a valuable asset for the broader scientific community.

The two scientific projects will combine a thorough molecular characterization of patients with different liver disease with studies on key and targetable pathways that drive key aspects of alcoholic hepatitis (AH) disease progression and outcome such as inflammation, injury and regeneration.

Project 1: ("Molecular Subtypes for Targeted Therapies in Liver disease") will identify molecular and cellular drivers of liver disease to provide a molecular classification using RNA sequencing, kinomic, metabolomic and novel systems biology approaches, and determine contributors to unfavorable outcomes and the associated progenitor cell accumulation.

Project 2: ("Determination of key drivers of the disease progression") The aim of the study is to describe histological, clinical and molecular characteristics that will make a particular disease evolve from early to advance form. We will use "omics" and novel systems, a biological approach as well as classic immunohistochemistry and histology stain technics. We will also use different imaging methodologies including second harmonic generation imaging microscopy (SHIM) and electronic microscopy to describe and identify specific histological patterns.

Project 3: Build a Human repository capable of providing a platform to develop projects 1 and 2.

ELIGIBILITY:
Patients with Alcoholic hepatitis:

* Inclusion:

  • Patients with a previous probable or possible AH episode will be defined following the guidelines proposed by the NIAAA.
* Exclusion

  * Terminal illness with less than 6 months live expectancy (e.g. advanced hepatocellular
  * carcinoma).
  * Patients who are pregnant or breastfeeding.
  * Complete portal vein thrombosis (PVT).
  * Previous liver transplant recipient

Patients with cirrhosis due to alcohol related liver disease without AH with or without a prior episode of decompensation.

* Inclusion:

  • Patients with a diagnosis of cirrhosis due to alcohol related liver disease according to clinical and/or analytic and/or radiological criteria.
* Exclusion

  * Terminal illness with less than 6 months live expectancy (e.g. advanced hepatocellular carcinoma).
  * Patients who are pregnant or breastfeeding.
  * Complete portal vein thrombosis
  * Previous liver transplant recipient
  * Current alcoholic hepatitis episode

Alcoholic liver disease with compensated never decompensated liver disease.

* Inclusion:

  * Patients diagnosed with an alcohol use disorder identification test (AUDIT) total scores of 8 or more OR Patients with a score lower than 8 in the AUDIT test but for whom there is a high suspicion of current or recent (within one year) AUD based on medical history, self reported history of excessive alcohol use, stigmata of alcohol use on physical exam, liver chemistry abnormalities, or alcohol induced organ involvement other than decompensated liver disease.
  * Patients who admit having a persistent alcohol intake of more than 40 g/daily for women and 60 g/daily for men.
  * Any stage of liver disease: from simple elevation of transaminases to any METAVIR or Ishack score assess by liver biopsy or by any validated noninvasive fibrosis score.
  * Patients without a preexistent liver fibrosis assessment for whom there is a high suspicion of liver disease according to clinical and/or analytic and/or radiological criteria will also be included.
* Exclusion

  * Patients with a past history of decompensated advanced liver disease (i.e. jaundice episodes, ascites, hepatic encephalopathy, variceal bleeding, hepatorenal syndrome) or known hepatocellular carcinoma.
  * Terminal illness with less than 6 months live expectancy (e.g. advanced hepatocellular carcinoma).
  * Patients who are pregnant or breastfeeding.

Non-Alcoholic Fatty Liver (NAFL)

* Inclusion:

  • Patients with a biopsy proven steatosis or steatosis and mild lobular inflammation OR Patients without a biopsy but with a high suspicious of NAFL and with at least three of the next 5 components of metabolic syndrome. (Waist circumference≥102/≥88 cm (40/35 inches) for men/women, Arterial pressure≥130/85mmHg or treated for hypertension, Fasting glucose 100mg/dl (5.6mmol/L) or treated for Type 2 diabetes, Serum triglyceride (triacylglycerols)>150mg/dL (>1.7mmol/L) if available, HDL cholesterol <40/50mg/dl for men/women (<1/<1.3 mmol/L) if available)
* Exclusion

  * Terminal illness with less than 6 months live expectancy (e.g. advanced hepatocellular carcinoma).
  * Patients who are pregnant or breastfeeding.
  * Complete portal vein thrombosis
  * Alcohol intake of more than 20g/daily.
  * Absence of other possible diagnoses (HCV and HBV negative, ANA's < 1:160, ASMA <1:80)

Patients with compensated early NASH.

* Inclusion:

  • Patients with a biopsy proven NASH and Metavir fibrosis score (or equivalent score) of F0-F2 OR Patients without a biopsy but with a high suspicious of NASH, with at least three of the next 5 components of metabolic syndrome and with a validated noninvasive score of F0-F2. (Waistcircumference≥102/≥88 cm (40/35 inches) for men/women, Arterial pressure≥130/85mmHg or treated for hypertension, Fasting glucose 100mg/dl (5.6mmol/L) or treated for Type 2 diabetes, Serum triglyceride (triacylglycerols) >150mg/dL (>1.7mmol/L) if available, HDL cholesterol <40/50mg/dl for men/women (<1/<1.3 mmol/L) if available)
* Exclusion

  * Terminal illness with less than 6 months live expectancy (e.g. advanced hepatocellular carcinoma).
  * Patients who are pregnant or breastfeeding.
  * Complete portal vein thrombosis.
  * Alcohol intake of more than 20g/daily.
  * Absence of other possible diagnoses (HCV and HBV negative, ANA's < 1:160, ASMA <1:80).
  * Decompensated liver diseases.

Patients with NASH advance fibrosis or cirrhosis compensated or decompensated.

* Inclusion:

  • Patients with a biopsyproven NASH and a METAVIR fibrosis score (or equivalent score) of F3-F4 OR Patients without a biopsy proven but with a high suspicious of NASH, with at least three of the next 5 components of metabolic syndrome and with a validated noninvasive fibrosis test score of F2-F3. (Waist circumference≥102/≥88 cm (40/35 inches) for men/women, Arterial pressure≥130/85mmHg or treated for hypertension, Fasting glucose 100mg/dl (5.6mmol/L) or treated for Type 2 diabetes, Serum triglyceride (triacylglycerols)>150mg/dL (>1.7mmol/L) if available, HDL cholesterol <40/50mg/dl for men/women (<1/<1.3 mmol/L) if available)
* Exclusion

  * Terminal illness with less than 6 months live expectancy (e.g. advanced hepatocellular carcinoma).
  * Patients who are pregnant or breastfeeding.
  * Complete portal vein thrombosis.
  * Alcohol intake of more than 20g/daily.
  * Absence of other possible diagnoses (HCV and HBV negative, ANA's < 1:160, ASMA < 1:80).

Dual NonAlcoholic Fatty Liver Disease and Alcoholic fatty liver disease (DAFLD) compensated or decompensated.

* Inclusion:

  * Patients diagnosed with an alcohol use disorder identification test (AUDIT) total scores of 8 or more or Patients with a score lower than 8 in the AUDIT test but for whom there is a high suspicion of current or recent (within one year) AUD based on medical history, self reported history of excessive alcohol use, stigmata of alcohol use on physical exam, liver chemistry abnormalities, or alcohol induced organ involvement other than decompensated liver disease.
  * Patients who admit having a persistent alcohol intake of more than 40 g/daily for women and 60 g/daily for men.
  * At least three of the next 5 components of metabolic syndrome (Waist circumference≥102/≥88 cm (40/35 inches) for men/women, Arterial pressure≥130/85mmHg or treated for hypertension, Fasting glucose 100mg/dl (5.6mmol/L) or treated Type 2 diabetes, Serum triglyceride (triacylglycerols)>150mg/dL (>1.7mmol/L), HDL <40/50mg/dl for men/women (<1/<1.3 mmol/L).)
  * BMI≥30
  * Any stage of liver disease: from simple elevation of transaminases to any METAVIR orIshack score assess by liver biopsy or by any validated noninvasive methods.
  * Patients without a preexistent liver fibrosis assessment for whom there is a high suspicion of liver disease according to clinical and/or analytic and/or radiological criteria will also be included.
* Exclusion

  * Terminal illness with less than 6 months live expectancy (e.g. advanced hepatocellular carcinoma).
  * Patients who are pregnant or breastfeeding.
  * Complete portal vein thrombosis.
  * Absence of other possible diagnoses (HCV and HBV negative, ANA's < 1:160, ASMA < 1:80).
  * A probable or possible episode of Alcoholic Hepatitis as defined by the NIAAA guidelines.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Alcoholic Steatohepatitis and Alcoholic liver disease
  2. Nonalcoholic fatty liver disease (NAFLD) and Nonalcoholic Steatohepatitis (NASH)
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Molecular Subtypes for Targeted Therapies in Liver disease | 5 years
  * Generation of consistent non-invasive molecular footprints of disease severity and prognosis: plasma and peripheral blood cells from groups of patients with different disease prognosis will be analyzed by means of high throughput proteomics (Mass Spectrometry and aptamer mediated identification) and single cell RNA sequencing, respectively. Data will be integrated with liver RNA-sequencing to detect relevant liver fingerprints in plasma.
  * Mechanisms of ductular reaction and hepatocyte de-differentiation will be studied by micro-dissection and region-specific RNA-sequencing.
  * Mechanisms of hepatocyte dedifferentiation will be evaluated using methylation bead chip and chromatin immunoprecipitation coupled to DNA sequencing (ChIP-seq) of histone marks related with activation, enhancement, poisoning and repression of gene expression.
Determination of key drivers of the disease progression | 5-10 years
  * To describe and identified the histological patters in each phase of the disease (using imaging technics, including second harmonic generation imaging microscopy and electronic microscopy as well as classical IHC technics)
  * To quantified and compare the degree of hepatic steatosis and fibrosis assessed by non-invasive techniques such as FibroScan® (CAP controlled attenuation parameter) across different cohorts of patients and across the different stages of the disease within the same patient's phenotype.
  * To identify the main genetic. psychosocial, and environmental factors influencing the development of advanced liver fibrosis among patients with known or suspected excessive alcohol intake. Through DNA
repository capable of providing a framework fro the other outcomes | 2-10 years
  To develop a bio-specimen bank comprised of plasma, DNA, and other biological specimens obtained from patients with alcoholic hepatitis, control disease and healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Jaideep Behari, MD, PhD, Principal Investigator — Associate Professor
Locations (1):
- University of Pittsburgh Medical center, Pittsburgh, Pennsylvania, United States